CLINICAL TRIAL: NCT00241670
Title: Fluorescence-guided Resection of Malignant Gliomas With 5-Aminolevulinic Acid (5-ALA) vs. Conventional Resection
Brief Title: Fluorescence-guided Resection of Malignant Gliomas With 5-Aminolevulinic Acid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: medac GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MC-ALS.3/GLI
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Brain Cancer; Brain Tumors; Cancer of Brain; Primary Brain Tumors; Brain Tumor, Primary
MeSH Terms: conditions — Brain Neoplasms | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 5-aminolevulinic acid (Experimental)
  Interventions: Drug: 5-aminolevulinic acid (5-ALA)
- Conventional resection (No Intervention)

INTERVENTIONS:
Drug: 5-aminolevulinic acid (5-ALA) — 1.5 grams 5-ALA dissolved in 50 ml water, single dose, orally, 2-4 hours prior to surgery
  Arms: 5-aminolevulinic acid

SUMMARY:
The aim of the study "Fluorescence-guided resection of malignant gliomas with 5-Aminolevulinic acid (5-ALA) vs. conventional resection" is to determine how accurately contrast agent-accumulating tumour can be removed by primary surgery and to assess the clinical usefulness of this method.

DETAILED DESCRIPTION:
Malignant gliomas are locally invasive tumors that carry a dismal prognosis despite a combination of surgery, radiotherapy and chemotherapy. Cytoreductive surgery is generally considered beneficial but complete resection of contrast enhancing tumor is achieved in less than 20 % of patients, one reason being the difficulty in discerning marginal, enhancing tumor intraoperatively.

Five-aminolevulinic acid (5-ALA) leads to the accumulation of fluorescent porphyrins in malignant gliomas, a phenomenon under exploration for intraoperative identification and resection of these tumors. This study investigated the benefit derived from fluorescent-guided resections using 5-ALA on surgical radicality, progression-free survival and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Radiological suspicion of a unilocular malignant glioma with distinct ring- or garland-shaped contrast agent-accumulating tumour structures and a core of reduced intensity in the MRI (central necroses) with no significant non-staining tumour tissue (exclusion of a secondary malignant glioma).
* Indication for surgical tumour resection. If radical resection is planned, the location of the contrast agent-accumulating tumour should allow complete resection.
* First operation of the tumour, no other tumour-specific pretreatment
* Karnofsky at least 70 %
* Patient's written informed consent
* Age 18-72 years

Exclusion Criteria:

* Tumour location in the midline, basal ganglia, cerebellum or brain stem
* More than one contrast agent-accumulating lesion unrelated to the primary tumour or extracerebral metastases
* Porphyria, hypersensitivity to porphyrins
* Renal insufficiency: Creatinine > 2.0 mg/dl
* Hepatic insufficiency: Bilirubin > 3 mg/dl
* Quick test < 60 %
* gamma-GT > 70 U/I
* Malignancies other than basaliomas
* Existing or planned pregnancy or lactation, or inadequate contraception
* Simultaneous participation in another clinical trial or participation in another clinical trial in the 30 days preceding randomisation

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 1999-10; Primary Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
1. Percentage of patients with a histologically confirmed malignant glioma (grade III or IV -WHO) without definite residual contrast agent-accumulating tumour in the early post-operative control MRI (within 72 hours of the operation). | Within 72 hours after surgery
2. Progression-free survival 6 months after primary surgical treatment of a malignant gli-oma in patients with histologically confirmed malignant glioma (grade III or IV -WHO). | Within 6 month after surgery

SECONDARY OUTCOMES:
1. Overall survival. | Until 18 months after surgery
2. Progression-free survival (PFS) 9, 12, 15 and 18 months after primary surgical treatment | Until 18 months after surgery
3. Volume of residual tumour | After surgery
4. Toxicity after oral administration of 5-Aminolevulinic acid. | Until 18 month after surgery
5. Neurological condition 7 days, 6 and 12 weeks, 6, 9, 12, and 18 months after primary surgical treatment | Until 18 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Juergen Reulen, MD, Study Chair — Ludwig-Maximilians - University of Munich

REFERENCES:
- [Derived] Stummer W, Pichlmeier U, Meinel T, Wiestler OD, Zanella F, Reulen HJ; ALA-Glioma Study Group. Fluorescence-guided surgery with 5-aminolevulinic acid for resection of malignant glioma: a randomised controlled multicentre phase III trial. Lancet Oncol. 2006 May;7(5):392-401. doi: 10.1016/S1470-2045(06)70665-9. PMID 16648043